CLINICAL TRIAL: NCT00389285
Title: A Phase 1/2, Open-Label, Dose Escalation Study to Assess the Safety and Pharmacokinetics of Recombinant Interleukin 21 (rIL-21) Administered Concomitantly With Sorafenib (Nexavar) in Subjects With Metastatic Renal Cell Carcinoma
Brief Title: Study of Recombinant Interleukin 21 in Combination With Sorafenib for Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Naomi Hunder, Medical Monitor, ZymoGenetics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 494F01
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Carcinoma, Renal Cell
Keywords: Carcinoma, renal cell; interleukin-21; sorafenib; Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

INTERVENTIONS:
Drug: rIL-21 only — Part 1: rIL-21, IV, Day 1-5 and 15-19 of each 6-week treatment course
Drug: rIL-21 + sorafenib — Part 2: rIL-21 IV, Day 1-5 and 15-19 of each 6-week treatment course + sorafenib (up to 400 mg taken orally twice daily)

SUMMARY:
The purpose of the study is to evaluate whether recombinant IL-21 used in combination with sorafenib is safe for patients with metastatic renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
This is a Phase 1/2 open-label dose-escalation study of rIL-21 given in combination with sorafenib to patients with metastatic RCC. The Phase 1 part of this study will estimate the maximum tolerated dose of rIL-21 given for 1 treatment course (consisting of two 5-day cycles of rIL-21) in combination with a standard dose of sorafenib administered during a 6-week treatment course. Increasing doses of rIL-21 will be studied sequentially in different groups of patients. The Phase 2 part of the study will further evaluate the safety and preliminary antitumor activity of rIL-21 at the dose recommended from Phase 1 in combination with sorafenib. Patients will be evaluated for safety over the course of the study. Disease evaluation (tumor restaging) will be performed during the last week of each 6-week treatment course. Patients with stable disease or better at this evaluation may go on to receive additional treatment courses. Patients may be in the study for 2 to 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RCC of predominantly clear cell histology
* Either no prior treatment or a maximum of 2 prior treatment regimens for metastatic RCC that included no more than 1 treatment regimen targeting the vascular endothelial growth factor (VEGF) pathway (Phase 1 only)
* At least 1 but no more than 2 prior systemic therapies for metastatic RCC that included no more than 1 therapy targeting the VEGF pathway (Phase 2 only)
* Disease measurable per the Response Evaluation Criteria in Solid Tumors (RECIST) (Phase 2 only)

Exclusion Criteria:

* Presence of acute infection or other significant systemic illness
* Central nervous system involvement by malignancy
* History of other cancer within 5 years
* Previously received rIL-21 or sorafenib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety profile, including incidence and severity of adverse events | During treatment and 28 days after last dose of rIL-21

SECONDARY OUTCOMES:
Objective response rate at recommended dose of rIL-21 | Every 6 weeks during treatment and then every 3 months after last dose of rIL-21 until 3 months after median survival is reached
Progression-free survival at recommended dose of rIL-21 | Every 6 weeks during treatment and then every 3 months after last dose of rIL-21 until 3 months after median survival is reached
Pharmacokinetic profiles of rIL-21 and sorafenib | rIL-21: During treatment and 15 days after dosing; sorafenib: During treatment and 22 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hunder, MD, Study Director — ZymoGenetics
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Derived] Bhatia S, Curti B, Ernstoff MS, Gordon M, Heath EI, Miller WH Jr, Puzanov I, Quinn DI, Flaig TW, VanVeldhuizen P, Byrnes-Blake K, Freeman JA, Bittner R, Hunder N, Souza S, Thompson JA. Recombinant interleukin-21 plus sorafenib for metastatic renal cell carcinoma: a phase 1/2 study. J Immunother Cancer. 2014 Jan 27;2:2. doi: 10.1186/2051-1426-2-2. eCollection 2014. PMID 24829759